CLINICAL TRIAL: NCT04569851
Title: Clinical Characteristics and Prognostic Factors of Patients With COVID-19 Using Big Data and Artificial Intelligence Techniques (BigCoviData)
Brief Title: Clinical Characteristics and Prognostic Factors of Patients With COVID-19 (Coronavirus Disease 2019)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Savana Research (Network)
Collaborators: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: BigCoviData
Record Dates: First submitted 2020-04-11; First posted 2020-09-30 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Infection
Keywords: Artificial Intelligence; Electronic health record; Intensive care unit; Natural language processing; Machine Learning; Real-world evidence; SARS-CoV-2 (Severe acute respiratory syndrome coronavirus 2); COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, non-interventional, retrospective study using data captured in the EHRs (Electronic Health Records) of the participating hospital sites to determine factors that predict disease prognosis and outcomes in COVID-19 patients, specifically: Hospitalization/Off-site monitoring, transfer to ICU and/or need for medical mechanical ventilation (both invasive and non- invasive), length of ICU stay, and outcome (cure/ hospital discharge, in-hospital death)

DETAILED DESCRIPTION:
Data captured in the EHRs will be collected from all available departments, including inpatient hospital, outpatient hospital, emergency room, etc. for virtually all types of provided services in each participating site. The study period will be from January 1, 2020 to the most recent data available.

* Primary objective To determine factors that predict disease prognosis and outcomes in COVID-19 patients, specifically: Hospitalization/Off-site monitoring, transfer to ICU and/or need for medical mechanical ventilation (both invasive and non- invasive), length of ICU stay, and outcome (cure/ hospital discharge, in-hospital death)
* Secondary objectives

  * To describe the demographic and clinical characteristics of COVID-19 patients
  * To describe the patient management (treatment and procedures) in the target population
  * To describe the outcomes of COVID-19 (discharge, hospitalization, transfer to ICU/ mechanical medical ventilation, in-hospital death) in relation to patients' clinical and demographic characteristics, and treatment received
  * To determine whether the factors that predict COVID-19 prognosis and outcome also apply to other types of pneumonia.
* Exploratory objectives One of the goals of this study is to configure the Big Data system to unravel any hidden variable/s (and their associations) that may offer novel clinical insights into COVID-19 management.

ELIGIBILITY:
Inclusion Criteria:

* All patients with suspected COVID-19 infection, as captured in the patients' EHRs of the participating sites.

Exclusion Criteria:

* Not suspected COVID-10 infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of all patients with suspected COVID-19 infection, as captured in the patients' EHRs of the participating sites.
  Among the suspected COVID-19 cases, we will determine the following:
  * Confirmed positive cases (i.e., all patients who tested positive for COVID-19 ).
  * Confirmed negative cases (i.e., all patients who tested negative for COVID-19)
  * Possible cases (i.e., all patients with suspected COVID-19 but no/pending test results) To determine the characteristics of the patients according to their clinical outcome, we will study both the confirmed positive cases and all possible classes (with no/pending laboratory results) subpopulations
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Factors that predict disease prognosis and outcomes in COVID-19 patients - Hospitalization | From 1st Jan 2020
  All variables and outcomes will be extracted from the free-text narratives available in patients' EHRs Hospitalization
  * Percentage of hospitalized patients at diagnosis
  * Percentage of hospitalized patients after diagnosis
  * Percentage of non-hospitalized patients
  * Percentage of patients admitted to the ICU Disease outcome: Cure/Hospital Discharge/In-hospital death
  * Percentage of patients who have been discharged
Factors that predict disease prognosis and outcomes in COVID-19 patients - ICU | From 1st Jan 2020
  Transfer to ICU and/or need for medical ventilation
  * Time (in days) from diagnosis to ICU admission
  * Time (in days) from the date of first symptom to ICU admission
  * Time (in days) from hospital admission to ICU admission (in hospitalized patients) Percentage of patients not admitted to the ICU Length of ICU stay
  * Length of ICU stay (mean duration in days across all patients)

SECONDARY OUTCOMES:
The demographic and clinical characteristics of COVID-19 patients | From 1st Jan 2020
  Gender (% of male patients; % of female patients)
The demographic and clinical characteristics of COVID-19 patients-Age at diagnosis | From 1st Jan 2020
  Age (in years) at diagnosis
The demographic and clinical characteristics of COVID-19 patients -Percentage of patients in each age range | From 1st Jan 2020
  Percentage of patients in each age range (<2; 2-4; 5-14; 15-29; 30-39; 40-49; 50-59; 60-69; 70-79; >= 80).
The demographic and clinical characteristics of COVID-19 patients with available PCR (Polymerase Chain Reaction) results | From 1st Jan 2020
  Percentage of patients with available PCR results (Positive; Negative; Unknown) Percentage of patients with available IgG (immunoglobulin G)/IgM (immunoglobulin M) results (Positive; Negative; Unknown) Percentage of patients using Alcohol/Tobacco/Other substances (Yes/No/Former user/Unknown
The demographic and clinical characteristics of COVID-19 patientsTime since first symptom until diagnosis | From 1st Jan 2020
  Time (in days) since first symptom until diagnosis
The demographic and clinical characteristics of COVID-19 patients - Physical examination | From 1st Jan 2020
  Physical examination
  * BMI
The demographic and clinical characteristics of COVID-19 patients - Physical examination of patients who are pregnant | From 1st Jan 2020
  Physical examination
  * Percentage of patients who are pregnant
The demographic and clinical characteristics of COVID-19 patients - Physical examination Temperature | From 1st Jan 2020
  Physical examination
  * Temperature (in degrees Celsius) - Percentage of patients within temperature ranges (in degrees Celsius) (<37, 37-38, >38)
The demographic and clinical characteristics of COVID-19 patients - Physical examination Heart rate (bmp) | From 1st Jan 2020
  Physical examination
  * Heart rate (bmp) - Percentage of patients within low/normal/high ranges of heart rate
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Hematology, Hemoglobin | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Hematology:
  Hemoglobin (g/dl)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Hematology, Hemoglobin II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Hematology:
  Hemoglobin n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Hematology, Red Blood Cells | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Hematology:
  Red Blood Cells (106/µl)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Hematology, Red Blood Cells II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Hematology:
  Red Blood Cells n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Hematology: Platelet, Leukocyte, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Hematology:
  Platelet count (103/mm3) Leukocyte count (103/mm3) Neutrophils (103/mm3) Lymphocytes (103/mm3) Monocytes (103/mm3) Eosinophils (103/mm3) Basophils (103/mm3)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Hematology: Platelet, Leukocyte, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Hematology:
  Platelet count n(%) Leukocyte count n(%) Neutrophils n(%) Lymphocytes n(%) Monocytes n(%) Eosinophils n(%) Basophils n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Hematology- INR (International Normalized Ratio) | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Hematology:
  INR n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Hematology- INR II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Hematology:
  INR
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Biochemistry: Glucose, Cholesterol, Triglycerides | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Biochemistry:
  Glucose (mg/dl) Total cholesterol (mg/dl) Triglycerides (mg/dl)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Biochemistry: Glucose, Cholesterol, Triglycerides II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Biochemistry:
  Glucose n(%) Total cholesterol n(%) Triglycerides n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Biochemistry: Bilirubin | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Biochemistry:
  Total bilirubin (g/dL)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Biochemistry: Bilirubin II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Biochemistry:
  Total bilirubin n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other Values: Creatinine, Glucose | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other values:
  Creatinine in urine (mg/dl) Glucose in urine (mg/dl)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other Values: Creatinine, Glucose II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other values:
  Creatinine in urine n(%) Glucose in urine n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other Values: Procalcitonin | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other values:
  Procalcitonin level will be reported" (PCT) ng/mL
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other test: PH (Potential Hydrogen), O2 Saturation, FIO2 (Fractional Inspired Oxigen), PAFI [Blood pressure of oxygen / inspired fraction of oxygen (PaO2/FiO2)] | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other tests:
  pH pH n(%) O2 saturation (%) O2 saturation n(%) FIO2 (%) FIO2 n(%) PAFI (%) PAFI n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other test: PH | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other tests:
  pH
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other test: PH II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other tests:
  PH n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other test: O2 saturation, FIO2, PAFI | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other tests:
  O2 saturation (%) FIO2 (%) PAFI (%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other test: O2 saturation, FIO2, PAFI II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other tests:
  O2 saturation n(%) FIO2 n(%) PAFI n(%)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other test: pCO2 (partial pressure of carbon dioxide), pO2 (partial pressure of oxygen) | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other tests:
  pCO2 (mmHg) pO2 (mmHg)
The demographic and clinical characteristics of COVID-19 patients - Laboratory values: Other test: pCO2, pO2 II | From 1st Jan 2020
  Physical examination. Laboratory values at diagnosis
  Other tests:
  pCO2 n(%) pO2 n(%)
The demographic and clinical characteristics of COVID-19 patients- Comorbidities, Medication, Symptoms | From 1st Jan 2020
  * Percentage of patients with family history of selected comorbidities
  * Percentage of patients with existing selected comorbidities at diagnosis: Cardiovascular disease, Hypertension, Ischemic stroke, Heart Disease (Cardiopathy), etc.
  * Percentage of patients with medication use/procedures prior to diagnosis. The following medications/treatments will be considered: ACEI (angiotensin converting enzyme inhibitors), ARB (angiotensin receptor blocker), Diuretics, Beta-blocker, etc.
  * Percentage of patients showing the following signs and symptoms at diagnosis: Cough, Fever, Dyspnoea, Respiratory crackles, Diarrhoea, etc.
  * Percentage of patients showing the following signs and symptoms after diagnosis: Thromboembolic Disorder, Venous thrombosis, Pulmonary thromboembolism, Upper gastrointestinal bleeding, etc.
The patient management (treatment and procedures) in the target population | From 1st Jan 2020
  Percentage of patients assigned to the following procedures after diagnosis: Chest x-ray, Ultrasonography of thorax,Ultrasonography of lung, High resolution computed tomography, Computer tomography of chest, Echocardiogram, EKG Percentage of patients assigned to the following treatments after diagnosis: Oxygen therapy (Oxygen administration by nasal cannula, Oxygen administration by Venturi mask, High concentration oxygen therapy), Prone position, Noninvasive ventilation, Invasive mechanical ventilation,Tracheotomy, Extubation of trachea.
  Percentage of patients (and mean duration of treatment in days) prescribed with the following pharmacological agents after diagnosis: Lopinavir + Ritonavir, Darunavir + Ritonavir, Darunavir + Cobicistat, IFN (Interferon)- β1b, Chloroquine, Hydroxychloroquine, Antibiotics, Acetylcysteine,Corticosteroids,Selective immunosuppressants, Cyclosporine, Remdesivir, Antithrombotic agents (anticoagulants), Inhibitors of platelet aggregation.
The outcomes of COVID-19 (discharge, hospitalization, transfer to ICU/ mechanical medical ventilation, in-hospital death) in correlation to patients' clinical and demographic characteristics, and treatment received | From 1st Jan 2020
  The outcomes of COVID-19 (discharge, hospitalization, transfer to ICU/ mechanical medical ventilation, in-hospital death) in correlation to patients' clinical and demographic characteristics, and treatment received
  * Percentage of patients with selected comorbidities (see complete list above) at diagnosis in each outcome group (ICU-no ICU; hospitalization-no hospitalization; discharge-no discharge; death-no death)
  * Percentage of patients showing selected sings and symptoms (see complete list above) at diagnosis in each outcome group (ICU-no ICU; hospitalization-no hospitalization; discharge-no discharge; death-no death)

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Izquierdo, MD, PhD, Study Chair — Hospital Universitario de Guadalajara; Joan B Soriano, MD, PhD, Study Chair — Hospital Universitario La Princesa; Julio Ancochea, MD, PhD, Study Chair — Hospital Universitario La Princesa
Locations (2):
- Spain (2):
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario La Princesa, Madrid